CLINICAL TRIAL: NCT07046754
Title: Patient Care Pathway and Factors Influencing Their Choice to Consult in the Emergency Department or an Out-of-Hours Care Service: A Comparative Study
Acronym: PSP-FICU
Status: Active, not recruiting | Type: Observational
Sponsor: Gwladys M'BOUNGOU (Other)
Responsible Party: Sponsor-Investigator, Gwladys M'BOUNGOU, Physician, Centre Hospitalier de Martigues
Organization: Centre Hospitalier de Martigues (Other)
Other Study IDs: 2024_02_RIPH3_Thèse Interne Dr
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2024-10

CONDITIONS: This Study is to Evaluate the Prevalence; Patients Consulting the Emergency Department for Reasons Relating to General Medicine
Keywords: Patient care pathway,; consultation at the Emergency Department; Permanent Care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- group of patients consulting the Emergency Department
  Interventions: Other: type of consultation
- group of patients consulting the permanent care service

INTERVENTIONS:
Other: type of consultation — urgence care, permance care
  Groups: group of patients consulting the Emergency Department

SUMMARY:
It focuses on the patient care pathway and the factors influencing their choice to seek consultation in the Emergency Department or Out-of-Hours Care Service for issues that fall under general medicine.

In France, emergency services are increasingly overcrowded, particularly with cases that should be handled by general practitioners. This strain on the healthcare system, caused by the saturation of emergency departments, has consequences on the quality of care for true emergencies.

This study aims to better understand who these users are and why they choose the Emergency Department over other care options.

DETAILED DESCRIPTION:
the saturation of Emergencies is explained by the constant increase in the number of visits, the reasons for this dynamic have been studied very little. Social security emphasizes that the characteristics of patients consulting there are poorly known.

Several theses in general medicine have dealt with the relevance of the use of SAU and the difficulties encountered in these structures, but none have dealt with this subject in the Martigues basin. Likewise, if several studies question doctors, none has yet questioned, in mirror image, patients in emergency rooms and an unscheduled care center.

To try to answer these unknowns, we propose to interview both patients consulting in the Emergency Department and in the City Medical Center for reasons relating to general medicine. This comparative study aims to determine and compare these two populations while identifying the factors influencing their choice of consultation location.

Our hypotheses:

* A significant proportion of patients consult the emergency room for non-urgent reasons, which could be taken care of by general medicine.
* Patients consult the Emergency Department or Permanent Care Center because the attending physician is not available.
* Patients consult the Emergency Department because they were not referred by a healthcare professional before going there.
* Patients come to the Emergency Department because it better corresponds to their way of consuming care. (Open 24 hours a day, easily accessible.) The target population of the study corresponds to adult patients consulting spontaneously and by their own means for a reason relating to general medicine, whether at the SAU of the Martigues Hospital Center or at the Escaillon Care Center.

To be included in the study, patients must meet the following criteria:

* Patients aged 18 and over
* Patients who have given oral consent
* Patients with rights covered by Social Security
* Patients able to understand French
* Patients consulting for any reason for consultation in general medicine

We have established a list of these reasons based on reading scientific literature and our experience in the practice of general medicine.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and over.
* Patients who have given oral consent.
* Patients with rights covered by Social Security.
* Patients able to understand French.

Exclusion Criteria:

* Minor patient.

  * Illiterate patient.
  * Patients who do not have social security rights.
  * Patient under guardianship or curatorship.
  * Patient deprived of liberty.
  * Patient under legal protection.
  * Patients admitted for consultation for the reasons below:
* Chest pain
* Limb fracture/deformity
* Major trauma
* Wound
* All vital emergencies: neurological, hemodynamic, respiratory.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients who consult the emergency room vs. permanent care in the city of Martigues
Sampling Method: Non-Probability Sample
Enrollment: 194 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
prevalence | one days
  proportion of patients consulting the Emergency Department for a reason relating to general medicine

CONTACTS AND LOCATIONS:
Overall Officials: Bouriche Bouriche, doctor, Study Director — Centre Hospitalier de Martigues
Locations (1):
- CH de Martigues, Martigues, Bouches du Rhone, France

IPD SHARING:
Plan to Share IPD: No